CLINICAL TRIAL: NCT04191850
Title: Comparison of the Analgesic Effect Between Ultrasound-Guided Serratus Anterior Plane Block and Intercostal Nerve Block After Single Port Video-Assisted Thoracoscopic Surgery in Primary Spontaneous Pneumothorax
Brief Title: Ultrasound-Guided Serratus Anterior Plane Block in Pneumothorax Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Saeyoung Kim, MD, PhD, Associate professor, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-12-012-001
Record Dates: First submitted 2019-12-04; First posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Analgesia; Postoperative Pain; Pneumothorax
MeSH Terms: conditions — Agnosia; Pain, Postoperative; Pneumothorax

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intercostal Nerve Block (Active Comparator): Intercostal Nerve Block was performed just before closing the surgical incision while looking directly at the affected intercostal space. 10ml of 0.375% ropivacaine was delivered evenly at anterior and posterior intercostal spaces from the port site.
  Interventions: Procedure: Single Port Video-Assisted Thoracoscopic Surgery
- Serratus Anterior Plane Block (Experimental): Serratus Anterior Plane Block was performed just before the start of surgery after anesthetic induction through ultrasound-guidance. 20ml of 0.375% ropivacaine was slowly injected between the fascia of serratus anterior and latissimus dorsi near 5th rib.
  Interventions: Procedure: Single Port Video-Assisted Thoracoscopic Surgery

INTERVENTIONS:
Procedure: Single Port Video-Assisted Thoracoscopic Surgery — Single Port Video-Assisted Thoracoscopic wedge resection was performed for primary spontaneous pneumothorax.

SUMMARY:
A prospective randomized controlled study was undertaken to compare the postoperative analgesic effect between ultrasound-guided serratus anterior plane block and intercostal nerve block after single port video-assisted thoracoscopic surgery with primary spontaneous pneumothorax.

DETAILED DESCRIPTION:
Post-thoracotomy pain is one of the most notorious postsurgical pains that one can experience. The pain is known to last for an extensive period of time with significantly high intensity.

In field of thoracic surgery, video-assisted thoracoscopic surgery has been played an important role in alleviating the postoperative pain. Furthermore, single-port thoracoscopic surgery, which reduces the number of surgical incision, is increasingly carried out by many institutions world widely.

In field of anesthesiology, various attempts to alleviate post-thoracotomy pain have been tried along advancement of thoracic surgical techniques. It began with postoperative medication of non-steroid anti-inflammatory drugs, opioids and progressed into implementations such as local analgesia, thoracic epidural block, paravertebral block, intercostal nerve block, interpleural block and serratus anterior plane block.

Many analgesic methods have been applied to alleviate postoperative pain in patients who have undergone thoracoscopic surgeries. However, there are no prospective randomized controlled studies between intercostal nerve block and serratus anterior plane block in single port video-assisted thoracoscopic surgeries. The main purpose of this study is to compare and analyze the effects between conventional intercostal nerve block and newly introduced serratus anterior plane block in primary spontaneous pneumothorax patients who have undergone single port video-assisted thoracoscopic wedge resection. This prospective study will discover the efficacy and differences between two methods.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) physical status 1 or 2
2. primary spontaneous pneumothorax
3. elective single port video-assisted thoracoscopic wedge resection of the lung.

Exclusion Criteria:

1. secondary spontaneous pneumothorax
2. reoperation in ipsilateral thorax
3. a history of drug allergy for analgesics
4. participants who have difficulty understanding the study protocol
5. refusal of participants

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain: numeric rating scale | 3 hours later operation
  Postoperative pain will be evaluated using a numeric rating scale (0 being no pain, 10 being worst pain imaginable)
Postoperative pain: numeric rating scale | 6 hours later operation
  Postoperative pain will be evaluated using a numeric rating scale (0 being no pain, 10 being worst pain imaginable)
Postoperative pain: numeric rating scale | 12 hours later operation
  Postoperative pain will be evaluated using a numeric rating scale (0 being no pain, 10 being worst pain imaginable)
Postoperative pain: numeric rating scale | After removal of chest tube
  Postoperative pain will be evaluated using a numeric rating scale (0 being no pain, 10 being worst pain imaginable)

SECONDARY OUTCOMES:
Number of analgesics consumption | through study completion, an average of 1 year
  If the participant has additional analgesic requirement postoperatively, ketorolac 30mg will be injected intravenously when numeric rating scale score is measured as 4-5, and fentanyl 50㎍ is injected when numeric rating scale score is over 6.
Amount of analgesics consumption | through study completion, an average of 1 year
  If the participant has additional analgesic requirement postoperatively, ketorolac 30mg will be injected intravenously when numeric rating scale score is measured as 4-5, and fentanyl 50㎍ is injected when numeric rating scale score is over 6.

CONTACTS AND LOCATIONS:
Overall Officials: Saeyoung Saeyoung, Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Kyungpook national university hospital, Daegu, South Korea